CLINICAL TRIAL: NCT02869958
Title: Digital Action Plan for Asthma Exacerbations (PANAME)
Brief Title: Digital Action Plan for Asthma Attacks
Acronym: PANAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: P140316
Record Dates: First submitted 2016-07-05; First posted 2016-08-17 (Estimated); Last update posted 2020-12-04 (Actual); Status verified 2020-12

CONDITIONS: Asthma
Keywords: Asthma; Exacerbation; Treatment; Internet; Emergency care
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1: Written action plan (Active Comparator): Written action plan
  Interventions: Other: Written action plan
- 2: Digital action plan (Experimental): Written action plan + Digital action plan for asthma exacerbations Digital action plan for asthma exacerbation available through an AppWeb and requiring a connected device such as a Smartphone or a tablet computer. The patient must connect and describe the situation to obtain the names, doses and dosing of the treatment his/her physician has recommended for him/her according to the level of severity of the exacerbation
  Interventions: Other: Digital action plan for asthma exacerbations + Written action plan

INTERVENTIONS:
Other: Digital action plan for asthma exacerbations + Written action plan — Digital action plan for asthma exacerbation available through an AppWeb and requiring a connected device such as a Smartphone or a tablet computer. The patient must connect and describe the situation to obtain the names, doses and dosing of the treatment his/her physician has recommended for him/her according to the level of severity of the exacerbation
  Other Names: Digital action plan for asthma exacerbations
  Arms: 2: Digital action plan
Other: Written action plan
  Arms: 1: Written action plan

SUMMARY:
It is recommended that patients with asthma owned a written action plan which must include the names, doses and dosing of the treatment they should take when acute respiratory symptoms occur.

Current written action plans must be short to be readily used (1 page) and, therefore, cannot fit all acute situations. Moreover, they may not be available where and when required.

The investigators sought that a digital action plan, available through Smartphone or tablet computer connected to the internet, could adequately provide suitable action plans according to the severity of the described exacerbation, and would be more easily available when useful.

The aim of the study is to study the effect of the use of a digital action plan for asthma exacerbation, on the frequency of unscheduled medical contacts (phone calls, visits to physicians or to emergency departments, hospitalizations) in children and in adults with asthma. The investigators hypothesized that the use of the digital action plan could reduce avoidable unscheduled visits due to mild or moderate exacerbations that could successfully be managed by the patient or his/her caregivers.

DETAILED DESCRIPTION:
Asthma is a frequent chronic disease (10% prevalence in children and 7% in adults) during which acute exacerbations can occur that require adequate treatment, usually by the patients and/or his/her caregivers. Despite action plan for asthma exacerbation being recommended by national and international guidelines, urgent medical contact and often Emergency Department visits remain frequent for asthma exacerbation.

Reasons for medical contact may be related to the inefficiency of the current Written Action Plan because of its stereotyped advice whatever the level of severity of the exacerbation, and because the patients might not have the paper with him/her where and when he/she needs it.

The investigators sought that new electronic technologies could solve these issues of inadequacy of content and availability of the Written Action Plan.

A program was built to provide sets of advices according to the severity of the exacerbation described by the patient using simple clinical descriptors included in the Global Initiative for Asthma (GINA), and weighted by the medication already used for the exacerbation. In this way the investigators feel that patients could be more confident in the appropriate treatment proposed by the algorithm. Second, the possibility to connect through portable electronic devices (Smartphone, tablet computer) make the action readily available as far as an internet connection is possible.

The Digital Action Plan is designed to treat asthma exacerbations of all levels of severity and advice to visit a doctor within few days or to go at once to an emergency department as appropriate as by the situation based on the patients' information. The investigators designed a randomized study to assess the effect of the Digital Action Plan on unscheduled urgent medical contacts (phone calls, visits to physicians or to emergency departments, hospitalizations) in children and in adults with asthma.

Methodology of the study A multicenter, controlled, randomized, open study, comparative on 2 parallel groups recruited in private practice and in hospitals within or outside the APHP consortium.

Both arms have the Written Action Plan respecting the current recommendations; the experimental arm has in addition the possibility to connect to the AppWeb to obtain advices from the Digital Action Plan.

The investigators hypothesized that the use of the digital action plan could reduce avoidable unscheduled visits due to mild or moderate exacerbations that could successfully be managed by the patient or his/her caregivers. In the long run, this kind of program could also become a tool for telemedicine Statistical analysis : about 80% of children and adult patients included will have a exacerbation during the follow-up year. The expected effect of the Digital Action Plan is a 20% (relative variation) decrease of the main outcome : in Written Action Plan group, frequency = 0.8, in Digital Action Plan group, frequency = 0.64 (20% i.e. 0.16 reduction of frequency). Moreover, the Written Action Plan has been shown to result in a 25% decrease of unscheduled visits for severe exacerbation (4); we therefore hypothesize that the supplemental reduction in unscheduled visits induced by the Digital Action Plan will be smaller than that of Written Action Plan despite the recording of moderate exacerbations in addition to severe exacerbations. . With this features, samples of N= 121 per group are necessary (80% power, bilateral alpha risk of 5%). With an expected attrition of about 15%, a total of 280 patients will be included. This target can be achieved with regard to the activity of participating centers.

Number of participating centers = 43

ELIGIBILITY:
Inclusion criteria :

* children from 6 to 12 years or adults aged between 18 and 60 years
* typical asthma with medical diagnosis
* severe exacerbation (requiring ≥ 3 days of oral corticosteroids) during the previous 12 months
* Internet connexion through a private (patient's or parents' patient's if child) smartphone and/or a tablet computer
* no use of a written actin plan within the last 1 year
* agreement to have phone calls or email contacts during the 1 year follow-up of the study
* informed consent given, signed consent
* affiliation to a social security

Exclusion criteria :

* atypical asthma: isolated cough, exercise respiratory discomfort
* other respiratory disease (cystic fibrosis, COPD, etc.)
* Severe heart disease (except high blood pressure)
* smoking > 15 pack-years
* asthma requiring regular oral corticosteroids treatment
* asthma requiring inhaled controller treatment administered via nebulizations performed at home
* no health insurance coverage
* sister or brother already included in this study (applies only to children)
* pregnancy and breastfeeding

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 280 (Actual)
Dates: Start 2016-11-03 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2020-04-29 (Actual)

PRIMARY OUTCOMES:
Number of visits or unscheduled medical contacts | during the 1 year follow-up
  Frequency of urgent medical recourses (composite criterion): visits or unscheduled medical contacts + Emergency Departments visits or hospitalizations, in both arms of randomization
Emergency Departments visits or hospitalizations | during the 1 year follow-up
  Frequency of urgent medical recourses (composite criterion): visits or unscheduled medical contacts + Emergency Departments visits or hospitalizations, in both arms of randomization

SECONDARY OUTCOMES:
Adherence to the Digital Action Plan = number of moderate to severe exacerbations entered in the AppWeb with respect to all moderate to severe exacerbations reported | during the 1 year follow-up
Adherence to the Written Action Plan (number of times Written Action Plan was used with respect to all moderate to severe exacerbations) | during the 1 year follow-up
qualitative evaluation of the Digital Action Plan: descriptive study using a questionnaire filled out in the arm using the AppWeb | at 1 year
number of unscheduled visits or medical contacts during the 1 year follow-up | during the 1 year follow-up
number of visits in Emergency Departments | during the 1 year follow-up
number of hospitalizations (>6 hours) | during the 1 year follow-up
number of school or working days missed | during the 1 year follow-up
number of scheduled medical | during the 1 year follow-up
Cumulative dose (in mg/kg) of oral corticosteroids during the 1 year follow-up | during the 1 year follow-up
assessment of the level of asthma control (GINA criteria) by a phone call | every 3 months, during the 1 year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Nicole BEYDON, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (2):
- France (2):
  - Hôpital Privé Armand Brillard, Nogent-sur-Marne
  - MulticEnter French study coordinate by AP-HP, Paris

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Beydon N, Taille C, Corvol H, Valcke J, Portal JJ, Plantier L, Mangiapan G, Perisson C, Aubertin G, Hadchouel A, Briend G, Guilleminault L, Neukirch C, Cros P, Appere de Vecchi C, Mahut B, Vicaut E, Delclaux C. Digital Action Plan (Web App) for Managing Asthma Exacerbations: Randomized Controlled Trial. J Med Internet Res. 2023 Jun 29;25:e41490. doi: 10.2196/41490. PMID 37255277